CLINICAL TRIAL: NCT03363113
Title: Outcome of Botulinum Toxin Treatment for Oromandibular Dystonia
Acronym: rétroBODOM
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CE_20150630_7_LSM
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Dystonia; Orofacial
MeSH Terms: conditions — Dystonia | interventions — Botulinum Toxins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Botulinum Toxins — Injection of botulinum toxin in the muscles affected by oromandibular dystonia

SUMMARY:
Symptoms of oromandibular dystonia can be alleviated by injections of botulinum toxin. The scope of this study is to describe the efficacy of this procedure, by a retrospective systematic review of patients medical charts

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from oromandibular dystonia
* Medical follow up in the Fondation Ophtalmologique Rothschild (Paris)
* Treatment by at least one session of botulinum toxin injection

Exclusion Criteria:

* Patient cannot assess symptoms improvement using a Likert scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by botulinum toxin injection for oromandibular dystonia in the Fondation Rothschild (Paris)
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
Clinical improvement score | Two months
  Likert scale for the assessment of the clinical improvement after treatment